CLINICAL TRIAL: NCT02666365
Title: Pharmacokinetic Comparison of Cefazolin Redosing Strategy for Surgical Prophylaxis. Bolus Dose vs Continuous Infusion
Brief Title: Continuous v Bolus Infusion of Cefazolin During Ventral Hernia Repair
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Investigator decided not to proceed.
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Kunal Karamchandani, Assistant Professor of Anesthesiology, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00003845
Record Dates: First submitted 2016-01-25; First posted 2016-01-28 (Estimated); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Surgical Site Infections
Keywords: anesthesia; surgical antimicrobial prophylaxis; surgical site infections
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bolus infusion of Cefazolin (Active Comparator): Subjects undergoing a ventral hernia repair in this arm of the study will receive the surgical prophylactic, cefazolin, in a bolus infusion
  Interventions: Procedure: Bolus infusion of Cefazolin
- Continuous Infusion of Cefazolin (Active Comparator): Subjects undergoing a ventral hernia repair in this arm of the study will receive the surgical prophylactic, cefazolin, in a continuous infusion
  Interventions: Procedure: Continuous infusion of Cefazolin

INTERVENTIONS:
Procedure: Bolus infusion of Cefazolin — Subjects in the bolus infusion arm of the study will receive bolus infusions of cefazolin throughout the surgical procedure
  Other Names: Bolus infusion
  Arms: Bolus infusion of Cefazolin
Procedure: Continuous infusion of Cefazolin — Subjects in the continuous infusion arm of the study will receive a continuous infusion of the cefazolin throughout the surgical procedure
  Other Names: Continuous infusion
  Arms: Continuous Infusion of Cefazolin

SUMMARY:
Patients undergoing an elective ventral hernia repair will be randomly assigned to receive either bolus infusion or continuous infusion of the cefazolin as the prophylactic antibiotic. The blood concentrations of unbound cefazolin would be measured in their blood samples and the levels compared within the two groups with respect to their minimal inhibitory concentration (MIC) value.

DETAILED DESCRIPTION:
Patients who will be undergoing elective ventral hernia repair will be potential candidates for this study. Once identified, the surgical team will approach the participant for consent and inclusion in the study. On the day of surgery, the subjects will be assigned to either the Bolus Group (CB) or Continuous Infusion Group (CI) according to a randomly generated assignment procedure. During the procedure, the dose of prophylactic Cefazolin will be given an hour before surgery and will be administered in accordance to group assignment. Subjects in the CB will receive bolus infusions of Cefazolin every 4 hours till the end of surgery. Subjects in the CI group will receive an initial bolus injection of Cefazolin followed by a continuous infusion till the closure of skin incision. Blood samples will be taken during surgery at t=0, 15, 30 and 60 minutes and every hour following till the end of surgery or 6 hours (whichever comes sooner)

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Elective open Ventral hernia repair in CDC class one (clean) cases
* Planned operative time greater than 4 Hours
* Planned routine administration of cefazolin for pre-op prophylaxis
* No history of MRSA

Exclusion Criteria:

* Patients unable to give informed consent
* Allergy to cephalosporins
* Pre-existing documented infection or ostomy (class II-IV wounds)
* Received cefazolin within 24 hours before surgery
* Creatinine clearance < 30 ml/min
* Upstaging of wound class intra-op that results in the administration of additional antibiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03 (Estimated); Primary Completion 2019-03 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Difference in Area Under Curve (AUC) of Cefazolin plasma concentration and minimum inhibitory concentration (MIC) in both treatment arms | First four hours
  After blood sample collection is completed samples will be analyzed for plasma concentrations of cefazolin. This concentration will be compared with the standard minimum inhibitory concentration of Cefazolin. It is expected that the difference between AUC and MIC in the continuous infusion group will be higher than the bolus infusion group during the first four hours of surgery.

SECONDARY OUTCOMES:
Difference in AUC of plasma concentration between the two regimens for the entire duration of surgery | Duration of surgery
  After blood sample collection is completed samples will be analyzed for plasma concentrations of cefazolin. This concentration will be compared with the standard minimum inhibitory concentration of Cefazolin. It is expected that the difference between AUC and MIC in the continuous infusion group will be higher than the bolus infusion group for the entire duration of surgery.
Total dose of cefazolin administered during the surgery | Duration of surgery
Total dose of cefazolin administered during the first 24 hours | 24 hours after the beginning of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Kunal Karamchandani, MD, Principal Investigator — Milton S. Hershey Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] MILES AA, MILES EM, BURKE J. The value and duration of defence reactions of the skin to the primary lodgement of bacteria. Br J Exp Pathol. 1957 Feb;38(1):79-96. No abstract available. PMID 13413084
- [Background] Lee FM, Trevino S, Kent-Street E, Sreeramoju P. Antimicrobial prophylaxis may not be the answer: Surgical site infections among patients receiving care per recommended guidelines. Am J Infect Control. 2013 Sep;41(9):799-802. doi: 10.1016/j.ajic.2012.11.021. Epub 2013 Mar 13. PMID 23489739
- [Background] Hawn MT, Vick CC, Richman J, Holman W, Deierhoi RJ, Graham LA, Henderson WG, Itani KM. Surgical site infection prevention: time to move beyond the surgical care improvement program. Ann Surg. 2011 Sep;254(3):494-9; discussion 499-501. doi: 10.1097/SLA.0b013e31822c6929. PMID 21817889
- [Background] Stulberg JJ, Delaney CP, Neuhauser DV, Aron DC, Fu P, Koroukian SM. Adherence to surgical care improvement project measures and the association with postoperative infections. JAMA. 2010 Jun 23;303(24):2479-85. doi: 10.1001/jama.2010.841. PMID 20571014
- [Background] Bratzler DW, Dellinger EP, Olsen KM, Perl TM, Auwaerter PG, Bolon MK, Fish DN, Napolitano LM, Sawyer RG, Slain D, Steinberg JP, Weinstein RA; American Society of Health-System Pharmacists (ASHP); Infectious Diseases Society of America (IDSA); Surgical Infection Society (SIS); Society for Healthcare Epidemiology of America (SHEA). Clinical practice guidelines for antimicrobial prophylaxis in surgery. Surg Infect (Larchmt). 2013 Feb;14(1):73-156. doi: 10.1089/sur.2013.9999. Epub 2013 Mar 5. No abstract available. PMID 23461695
- [Background] Adembri C, Ristori R, Chelazzi C, Arrigucci S, Cassetta MI, De Gaudio AR, Novelli A. Cefazolin bolus and continuous administration for elective cardiac surgery: improved pharmacokinetic and pharmacodynamic parameters. J Thorac Cardiovasc Surg. 2010 Aug;140(2):471-5. doi: 10.1016/j.jtcvs.2010.03.038. Epub 2010 Jun 8. PMID 20570290
- [Background] Trent Magruder J, Grimm JC, Dungan SP, Shah AS, Crow JR, Shoulders BR, Lester L, Barodka V. Continuous Intraoperative Cefazolin Infusion May Reduce Surgical Site Infections During Cardiac Surgical Procedures: A Propensity-Matched Analysis. J Cardiothorac Vasc Anesth. 2015 Dec;29(6):1582-7. doi: 10.1053/j.jvca.2015.03.026. Epub 2015 Mar 31. PMID 26275516
- [Background] Ferraz AA, Siqueira LT, Campos JM, Araujo GC, Martins Filho ED, Ferraz EM. ANTIBIOTIC PROPHYLAXIS IN BARIATRIC SURGERY: a continuous infusion of cefazolin versus ampicillin/sulbactam and ertapenem. Arq Gastroenterol. 2015 Apr-Jun;52(2):83-7. doi: 10.1590/S0004-28032015000200002. PMID 26039823
- [Background] Finan KR, Vick CC, Kiefe CI, Neumayer L, Hawn MT. Predictors of wound infection in ventral hernia repair. Am J Surg. 2005 Nov;190(5):676-81. doi: 10.1016/j.amjsurg.2005.06.041. PMID 16226938
- [Background] Dunne JR, Malone DL, Tracy JK, Napolitano LM. Abdominal wall hernias: risk factors for infection and resource utilization. J Surg Res. 2003 May 1;111(1):78-84. doi: 10.1016/s0022-4804(03)00077-5. PMID 12842451
- [Background] Houck JP, Rypins EB, Sarfeh IJ, Juler GL, Shimoda KJ. Repair of incisional hernia. Surg Gynecol Obstet. 1989 Nov;169(5):397-9. PMID 2530641
- [Background] Kaafarani HM, Kaufman D, Reda D, Itani KM. Predictors of surgical site infection in laparoscopic and open ventral incisional herniorrhaphy. J Surg Res. 2010 Oct;163(2):229-34. doi: 10.1016/j.jss.2010.03.019. Epub 2010 Apr 1. PMID 20605590
- [Background] Blatnik JA, Krpata DM, Novitsky YW, Rosen MJ. Does a history of wound infection predict postoperative surgical site infection after ventral hernia repair? Am J Surg. 2012 Mar;203(3):370-4; discussion 374. doi: 10.1016/j.amjsurg.2011.12.001. PMID 22364903
- [Background] Buijk SE, Gyssens IC, Mouton JW, Metselaar HJ, Groenland TH, Verbrugh HA, Bruining HA. Perioperative pharmacokinetics of cefotaxime in serum and bile during continuous and intermittent infusion in liver transplant patients. J Antimicrob Chemother. 2004 Jul;54(1):199-205. doi: 10.1093/jac/dkh268. Epub 2004 Jun 2. PMID 15175266